CLINICAL TRIAL: NCT03642509
Title: Left Atrial Appendage Occlusion Versus Novel Oral Anticoagulation for Stroke Prevention in Atrial Fibrillation. A Multicenter Randomized Clinical Trial. (Occlusion-AF)
Brief Title: Left Atrial Appendage Occlusion Versus Novel Oral Anticoagulation for Stroke Prevention in Atrial Fibrillation
Acronym: Occlusion-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); Haukeland University Hospital (Other); Helsinki University Central Hospital (Other); Gødstrup Hospital (Other); Lund University Hospital (Other); Oslo University Hospital (Other); Trondheim University Hospital (Other); Rigshospitalet, Denmark (Other); Jena University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Occlusion-AF-AUH250418-32
Record Dates: First submitted 2018-07-06; First posted 2018-08-22 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Left atrial appendage occlusion; Novel oral anticoagulation
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Left Atrial Appendage Closure; N(4)-oleylcytosine arabinoside; edoxaban; apixaban; Rivaroxaban; Dabigatran

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open-label study with blinded outcome assessment by an independent clinical event committee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAAO group (Experimental): Patients will be treated with transcatheter left atrial appendage occlusion. The LAAO may be performed with the Amulet or Watchman device.
  Interventions: Device: Left atrial appendage occlusion
- NOAC group (Experimental): Patients will be treated with one of the currently available NOAC drugs; Apixaban, Dabigatran, Edoxaban or Rivaroxaban.
  Interventions: Drug: NOAC

INTERVENTIONS:
Device: Left atrial appendage occlusion — Interventional left atrial appendage occlusion with the Amulet or Watchman device
  Other Names: Left atrial appendage closure
  Arms: LAAO group
Drug: NOAC — Medical treatment arm. Patients will be treated with one of the available NOAC drugs; Apixaban, Dabigatran, Edoxaban or Rivaroxaban. The specific drug and dose is at the discretion of the treating physician.
  Other Names: Edoxaban; Apixaban; Rivaroxaban; Dabigatran
  Arms: NOAC group

SUMMARY:
Atrial fibrillation (AF) is progressively common, and increases the risk of stroke five-fold. Oral anticoagulation is the mainstay therapy; however, it increases the risk of bleeding. Moreover, 30% with AF and at risk of stroke are not in relevant anticoagulation. The randomized PROTECT-AF trial has demonstrated the superiority of left atrial appendage occlusion (LAAO) as compared to warfarin for prevention of the combined endpoint of stroke, major bleeding and cardiovascular mortality. However, studies comparing LAAO to therapy with novel oral anticoagulants (NOAC) have not been carried out.

This study aims to assess the effect of left atrial appendage occlusion (LAAO) to reduce the incidence of stroke, systemic embolism, major bleeding and all-cause mortality in patients with atrial fibrillation (AF) and a prior ischemic stroke or transient ischemic attack (TIA).

DETAILED DESCRIPTION:
An investigator-initiated multicenter, randomized open-label non-inferiority trial with blinded outcome evaluation (PROBE design). The active comparison LAAO is tested against NOAC therapy in a 1:1 stratified randomization. Patients should have AF, and an ischemic stroke or TIA within 6 months prior to enrollment. In total 750 patients will be included. Follow-up will be based on in-office and telephone follow-up during the first 3 years after randomization, along with up to 10 years long-term follow-up through the National Patient Registries.

The main study outcomes: The primary outcome is a composite of stroke (hemorrhagic or ischemic), systemic embolism, major bleeding or all-cause mortality assessed after at least two years follow-up for the last enrolled patient. Secondary outcomes will examine early and late safety outcome measures. The long-term outcome will be assessed up to 10-years after randomization through the National Patient Registries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* documented non-valvular atrial fibrillation (paroxysmal, persistent or permanent)
* Eligible for long-term Novel Oral Anticoagulation (NOAC) therapy
* Ischemic stroke within the recent 6 months verified by neuroimaging, or
* Transient ischemic attack within 6 months with proven cerebral ischemia based on cerebral magnetic resonance imaging (MRI)

Exclusion Criteria:

* Modified rankin scale > 3 at time of enrollment
* Glomerular filtration rate (GFR) below 15 ml/min/1.73 m2
* Contraindication towards long-term aspirin therapy
* Planned combined cardiovascular interventional procedures at the time of enrollment
* Terminal illness or cancer with life expectancy less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of stroke (ischemic and hemorrhagic), systemic embolism, major bleeding and all-cause mortality. | Up to 5-years from randomization
  The primary endpoint is the combined rate of stroke, systemic embolism, major bleeding and all-cause mortality.

SECONDARY OUTCOMES:
Incidence of ischemic stroke | 2-, 3-, 5- and 10-years
  The occurrence of an acute onset of a focal neurological deficit of presumed vascular origin lasting for ≥ 24 hours or resulting in death. Stroke is categorized as ischemic based on computed tomography (CT) or magnetic resonance imaging (MRI) of the brain or autopsy.
Incidence of hemorrhagic stroke | 2-, 3-, 5- and 10-years
  The occurrence of an acute onset of a focal neurological deficit of presumed vascular origin lasting for ≥ 24 hours or resulting in death. Stroke is categorized as hemorrhagic based on computed tomography (CT) or magnetic resonance imaging (MRI) of the brain or autopsy.
Incidence of systemic embolism | 2-, 3-, 5- and 10-years
  The occurrence of an acute vascular insufficiency or occlusion of the extremities or any non-CNS organ associated with clinical, imaging, surgical or autopsy evidence of arterial occlusion in the absence of other likely mechanism (e.g. trauma, atherosclerosis, or instrumentation).
Incidence of major or life-threatening bleeding | 2-, 3-, 5- and 10-years
  The occurrence of an overt bleeding associated with one or more of the following: decrease in hemoglobin of at least 3.0 g/dL, transfusion of 2 or more units of blood, causing hospitalization, requiring surgery, causing discontinuation of all antithrombotic therapy or pericardial bleeding with/without tamponade or occurring during the index LAAO procedure or during hospitalization for the index procedure (major bleeding). Life-threatening bleeding is defined as fatal bleeding, causing hypovolaemic shock or severe hypotension requiring vasopressor therapy or intervention, symptomatic bleeding in a critical organ (intracranial, intraspinal, intraocular, intramuscular with compartment syndrome, pericardial bleeding after hospitalization for the index LAAO) or overt bleeding with decrease in hemoglobin ≥ 5 g/dL or requiring transfusion of ≥ 4 units of blood.
Incidence of all-cause mortality | 2-, 3-, 5- and 10-years
  The occurrence of death from any cause
Incidence of Transient ischemic attack (TIA) | 2-, 3-, 5- and 10-years
  an episode of neurological dysfunction caused by focal brain, spinal cord or retinal ischemia leading to symptoms lasting less than 24 hours, without acute infarction based on neuroimaging.
Number of patients with a device-related complication | 2 months
  A complication related to the presence of the device. Device-related complications include:
  * Device embolization
  * Device erosion
  * Clinically significant device interference with surrounding structures. This includes structures at the implant location (circumflex coronary artery, mitral valve, pulmonary artery, pulmonary vein) or cardiovascular structures in the vicinity of the location to which the device migrated (if applicable).
  * Device thrombus
  * Device fracture
  * Device infection/endocarditis/pericarditis
  * Device perforation/laceration
  * Device allergy
Number of patients with a procedure-related complication | 2 months
  All complications related to the LAAO-procedure will be assessed.
Number of patients with a device success | 2 months
  Device deployed and implanted in correct position
Number of patients with technical success | 2 Months
  Exclusion of the left atrial appendage (LAA) achieved without device-related complications and no leak >5 mm on color Doppler TEE.
Number of patients with procedural success | 2 months
  Technical success and no procedure-related complications, except uncomplicated device embolization (i.e. device embolization resolved by percutaneous retrieval during the procedure without surgical intervention or damage to surrounding cardiovascular structures).
Number of patients with peri-device leaks at follow-up imaging | 2 months
  Detection of any peri-device flow/gap at follow-up cardiac CT/TEE.
Changes in functional status based on Modified Rankin Scale | 24 months
  The Modified Rankin scale is used to measure the degree of disability or dependence in daily activities caused by a stroke. The scale runs from 0-6, from no symptoms (0) to death (6).
Changes in Quality of life | 12 months
  Based on patient self-reported EuroQol-5D questionnaires. The EuroQol-5D is a standardized instrument to measure health-related quality of life. It includes five self-rated dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The questionnaire have 3 levels of severity for each of the five dimensions. It also includes a visual scale from 0 (worst thinkable health condition) to 100 (best thinkable health condition) to report an overall measure.
Compliance to NOAC | 2-, 3-, 5-, and 10-years
  Adherence to assigned NOAC therapy will be assessed through the National Prescription Registries.
Changes in neurological status based on National Institute of Health (NIH) Stroke scale score | 12 months
  Assessed by the NIH stroke scale at baseline and 12 month follow-up. A scale to quantify the neurological impairment caused by a stroke. It includes 11 items, each of which scores a specific ability between 0 to 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores are summed to calculate the total NIH Stroke Scale score, that can range from 0 to 42, with 0 being no symptoms.
  * Score 0: No stroke symptoms
  * Score 1-4: Minor stroke
  * Score 5-15: Moderate stroke
  * Score 16-20: Moderate to severe stroke
  * Score 21-42: Severe stroke

OTHER OUTCOMES:
Minor bleeding | 24 months
  Any bleeding clinically mentionable that does not qualify as life-threatening, disabling or major.
Comparison of the cost-effectiveness of LAAO and NOAC therapy | 24 months
  All costs and cost-effectiveness will be evaluated and compared between the two diagnostic strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Korsholm, MD, Study Chair — Aarhus University Hospital; Jens Erik Nielsen-Kudsk, MD DMSc Prof, Study Chair — Aarhus University Hospital; Dorte Damgaard, MD PhD, Study Chair — Aarhus University Hospital; Søren Paaske Johnsen, MD PhD Prof, Study Chair — Aalborg University Hospital
Locations (15):
- Denmark (5):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Odense University Hospital, Odense, Region Syddanmark
  - Aalborg University Hospital, Aalborg, The North Denmark Region
  - Rigshospitalet, Copenhagen
  - Regional Hospital West Jutland, Holstebro
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku
- Jena University Hospital, Jena, Germany
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - Trondheim University Hospital, Trondheim
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skånes University Hospital, Lund
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zoni-Berisso M, Lercari F, Carazza T, Domenicucci S. Epidemiology of atrial fibrillation: European perspective. Clin Epidemiol. 2014 Jun 16;6:213-20. doi: 10.2147/CLEP.S47385. eCollection 2014. PMID 24966695
- [Background] Marini C, De Santis F, Sacco S, Russo T, Olivieri L, Totaro R, Carolei A. Contribution of atrial fibrillation to incidence and outcome of ischemic stroke: results from a population-based study. Stroke. 2005 Jun;36(6):1115-9. doi: 10.1161/01.STR.0000166053.83476.4a. Epub 2005 May 5. PMID 15879330
- [Background] Blackshear JL, Odell JA. Appendage obliteration to reduce stroke in cardiac surgical patients with atrial fibrillation. Ann Thorac Surg. 1996 Feb;61(2):755-9. doi: 10.1016/0003-4975(95)00887-X. PMID 8572814
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Diener HC, Connolly SJ, Ezekowitz MD, Wallentin L, Reilly PA, Yang S, Xavier D, Di Pasquale G, Yusuf S; RE-LY study group. Dabigatran compared with warfarin in patients with atrial fibrillation and previous transient ischaemic attack or stroke: a subgroup analysis of the RE-LY trial. Lancet Neurol. 2010 Dec;9(12):1157-1163. doi: 10.1016/S1474-4422(10)70274-X. Epub 2010 Nov 6. PMID 21059484
- [Background] Hankey GJ, Patel MR, Stevens SR, Becker RC, Breithardt G, Carolei A, Diener HC, Donnan GA, Halperin JL, Mahaffey KW, Mas JL, Massaro A, Norrving B, Nessel CC, Paolini JF, Roine RO, Singer DE, Wong L, Califf RM, Fox KA, Hacke W; ROCKET AF Steering Committee Investigators. Rivaroxaban compared with warfarin in patients with atrial fibrillation and previous stroke or transient ischaemic attack: a subgroup analysis of ROCKET AF. Lancet Neurol. 2012 Apr;11(4):315-22. doi: 10.1016/S1474-4422(12)70042-X. Epub 2012 Mar 7. PMID 22402056
- [Background] Easton JD, Lopes RD, Bahit MC, Wojdyla DM, Granger CB, Wallentin L, Alings M, Goto S, Lewis BS, Rosenqvist M, Hanna M, Mohan P, Alexander JH, Diener HC; ARISTOTLE Committees and Investigators. Apixaban compared with warfarin in patients with atrial fibrillation and previous stroke or transient ischaemic attack: a subgroup analysis of the ARISTOTLE trial. Lancet Neurol. 2012 Jun;11(6):503-11. doi: 10.1016/S1474-4422(12)70092-3. Epub 2012 May 8. PMID 22572202
- [Background] Rost NS, Giugliano RP, Ruff CT, Murphy SA, Crompton AE, Norden AD, Silverman S, Singhal AB, Nicolau JC, SomaRaju B, Mercuri MF, Antman EM, Braunwald E; ENGAGE AF-TIMI 48 Investigators. Outcomes With Edoxaban Versus Warfarin in Patients With Previous Cerebrovascular Events: Findings From ENGAGE AF-TIMI 48 (Effective Anticoagulation With Factor Xa Next Generation in Atrial Fibrillation-Thrombolysis in Myocardial Infarction 48). Stroke. 2016 Aug;47(8):2075-82. doi: 10.1161/STROKEAHA.116.013540. Epub 2016 Jul 7. PMID 27387994
- [Background] Gadsboll K, Staerk L, Fosbol EL, Sindet-Pedersen C, Gundlund A, Lip GYH, Gislason GH, Olesen JB. Increased use of oral anticoagulants in patients with atrial fibrillation: temporal trends from 2005 to 2015 in Denmark. Eur Heart J. 2017 Mar 21;38(12):899-906. doi: 10.1093/eurheartj/ehw658. PMID 28110293
- [Background] Hellfritzsch M, Husted SE, Grove EL, Rasmussen L, Poulsen BK, Johnsen SP, Hallas J, Pottegard A. Treatment Changes among Users of Non-Vitamin K Antagonist Oral Anticoagulants in Atrial Fibrillation. Basic Clin Pharmacol Toxicol. 2017 Feb;120(2):187-194. doi: 10.1111/bcpt.12664. Epub 2016 Oct 28. PMID 27580086
- [Background] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Background] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Background] Reddy VY, Doshi SK, Kar S, Gibson DN, Price MJ, Huber K, Horton RP, Buchbinder M, Neuzil P, Gordon NT, Holmes DR Jr; PREVAIL and PROTECT AF Investigators. 5-Year Outcomes After Left Atrial Appendage Closure: From the PREVAIL and PROTECT AF Trials. J Am Coll Cardiol. 2017 Dec 19;70(24):2964-2975. doi: 10.1016/j.jacc.2017.10.021. Epub 2017 Nov 4. PMID 29103847
- [Background] Boersma LV, Schmidt B, Betts TR, Sievert H, Tamburino C, Teiger E, Pokushalov E, Kische S, Schmitz T, Stein KM, Bergmann MW; EWOLUTION investigators. Implant success and safety of left atrial appendage closure with the WATCHMAN device: peri-procedural outcomes from the EWOLUTION registry. Eur Heart J. 2016 Aug;37(31):2465-74. doi: 10.1093/eurheartj/ehv730. Epub 2016 Jan 27. PMID 26822918
- [Background] Tzikas A, Shakir S, Gafoor S, Omran H, Berti S, Santoro G, Kefer J, Landmesser U, Nielsen-Kudsk JE, Cruz-Gonzalez I, Sievert H, Tichelbacker T, Kanagaratnam P, Nietlispach F, Aminian A, Kasch F, Freixa X, Danna P, Rezzaghi M, Vermeersch P, Stock F, Stolcova M, Costa M, Ibrahim R, Schillinger W, Meier B, Park JW. Left atrial appendage occlusion for stroke prevention in atrial fibrillation: multicentre experience with the AMPLATZER Cardiac Plug. EuroIntervention. 2016 Feb;11(10):1170-9. doi: 10.4244/EIJY15M01_06. PMID 25604089
- [Background] Landmesser U, Schmidt B, Nielsen-Kudsk JE, Lam SCC, Park JW, Tarantini G, Cruz-Gonzalez I, Geist V, Della Bella P, Colombo A, Zeus T, Omran H, Piorkowski C, Lund J, Tondo C, Hildick-Smith D. Left atrial appendage occlusion with the AMPLATZER Amulet device: periprocedural and early clinical/echocardiographic data from a global prospective observational study. EuroIntervention. 2017 Sep 20;13(7):867-876. doi: 10.4244/EIJ-D-17-00493. PMID 28649053
- [Background] Sahay S, Nombela-Franco L, Rodes-Cabau J, Jimenez-Quevedo P, Salinas P, Biagioni C, Nunez-Gil I, Gonzalo N, de Agustin JA, Del Trigo M, Perez de Isla L, Fernandez-Ortiz A, Escaned J, Macaya C. Efficacy and safety of left atrial appendage closure versus medical treatment in atrial fibrillation: a network meta-analysis from randomised trials. Heart. 2017 Jan 15;103(2):139-147. doi: 10.1136/heartjnl-2016-309782. Epub 2016 Sep 1. PMID 27587437
- [Background] Tzikas A, Holmes DR Jr, Gafoor S, Ruiz CE, Blomstrom-Lundqvist C, Diener HC, Cappato R, Kar S, Lee RJ, Byrne RA, Ibrahim R, Lakkireddy D, Soliman OI, Nabauer M, Schneider S, Brachman J, Saver JL, Tiemann K, Sievert H, Camm AJ, Lewalter T. Percutaneous left atrial appendage occlusion: the Munich consensus document on definitions, endpoints and data collection requirements for clinical studies. EuroIntervention. 2016 May 17;12(1):103-11. doi: 10.4244/EIJV12I1A18. PMID 27173870